CLINICAL TRIAL: NCT03768687
Title: A Real-world Study of on Albumin-bound Paclitaxel as First-line Treatment of Patients With Non-operative Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: A Real-world Study of Albumin-bound Paclitaxel in the Treatment of Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Baorui Liu, chief doctor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: EXPLORE-PC101
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; albumin-bound paclitaxel
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients enrolled in the study underwent whole-gene sequencing based on their willingness to take tumor tissue samples and blood samples.All samples need tissue samples and peripheral blood as control. Tissue samples can be wax blocks, fresh surgical tissues,tissues through puncture biopsy, laparoscopic biopsy and other biopsy. Sampling should be conducted within 1 week before enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pancreatic cancer progresses rapidly and has a higher death rate. Albumin-bound paclitaxel is a new generation of paclitaxel . Albumin-bound paclitaxel is recommended as a class 1A evidence treating patients with pancreatic cancer.The purpose of this study was to further observe and evaluate the clinical efficacy and safety of albumin-bound paclitaxel in the treatment of non-operative locally advanced or metastatic pancreatic cancer and to explore the prognostic factors .

DETAILED DESCRIPTION:
This is a prospective, single-arm, observational study. After the subjects meet the inclusive and exclusive criteria, then they will receive albumin-bound paclitaxel treatment. The researchers can choose the treatment based on albumin-bound paclitaxel and choose dosage according to the patient's condition.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 -80, male or female;
2. Non-operative patients with locally advanced or metastatic pancreatic cancer diagnosed by pathology or histology (except islet cell carcinoma);
3. The patient has not received standard systematic treatment in the past, and the metastatic site has not received any local treatment, including radiotherapy, chemotherapy, surgical treatment, etc.;
4. At least one measurable lesion (CT scan length of tumor lesion is greater than 10 mm, CT scan short diameter of lymph node lesion is greater than 15 mm, scanning layer thickness is not greater than 5 mm);
5. The subjects volunteered to participate in this study and signed the informed consent form, with good compliance to follow-up.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Patients allergy to albumin-bound paclitaxel or its excipients
3. Patients with albumin-bound paclitaxel contraindication;
4. Doctors consider those who are not suitable for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-12-20 (Estimated); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 3 weeks
  the date from enrollment to the first occurrence of disease progression or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Baorui Liu, Doctor, Principal Investigator — The Affiliated Hospital of Nanjing University Medical School
Locations (1):
- The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dai W, Qiu X, Lu C, Zou Z, Sha H, Kong W, Liu B, Du J. AGIG Chemo-Immunotherapy in Patients With Advanced Pancreatic Cancer: A Single-Arm, Single-Center, Phase 2 Study. Front Oncol. 2021 Oct 13;11:693386. doi: 10.3389/fonc.2021.693386. eCollection 2021. PMID 34722242